CLINICAL TRIAL: NCT06753292
Title: The Influence of Combining the Pulmonary Recruitment Maneuver with Active Gas Aspiration on Post-laparoscopic Shoulder Pain in Patients Having a Gynecologic Laparoscopy, Randomized Double Blinded Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Essam Salama Hammam, resident doctor at Assiut University hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: pulm recruit gas aspir Gyn lap
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Post Laparoscopic Shoulder Pain
Keywords: pulmonary recruitment maneuver; active gas aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group 1 (Experimental): The surgeon will be instructed to actively aspirate the intraperitoneal CO2 gas
  Interventions: Procedure: active gas aspiration
- group 2 (Experimental): The surgeon will be instructed to apply PRM pressures. patients will receive the PRM which consisted of five manual pulmonary inflations,
  Interventions: Procedure: pulmonary recruitment maneuver

INTERVENTIONS:
Procedure: active gas aspiration — surgeon will be instructed to actively aspirate the intraperitoneal CO2 gas
  Arms: group 1
Procedure: pulmonary recruitment maneuver — patients will receive the PRM which consisted of five manual pulmonary inflations, where each positive pressure inflation will be done for 5 s at a maximum pressure of 30 cm H2O, manually by using the APL valve in the anesthesia machine. The patient will be in a Trendelenburg position (30°). The fifth positive pressure inflation lasted for approximately 5 s. During that time, the patient will be closely monitored, while the anesthesiologist performed PRM
  Arms: group 2

SUMMARY:
Laparoscopy is among the most used minimally invasive procedures that can reduce postoperative pain, lessen the duration of hospital stay and facilitate recovery. Laparoscopy has been widely used in various abdominal surgeries, such as gastrectomy, cholecystectomy, appendectomy, hernia and gynecological surgery . However, the post-laparoscopic shoulder pain (PLSP) often occurs following laparoscopic surgeries, and its reported incidence varies from 35-80% This study aims to assess the effect of combining pulmonary recruitment maneuvers (PRM) with active gas aspiration on post-laparoscopic shoulder pain in patients undergoing gynecological laparoscopic procedures.

DETAILED DESCRIPTION:
The PLSP can even remain for up to three days and often upsets the patients . Moreover, it can increase the costs of healthcare owing to an increased usage of analgesics, delayed discharge, and even re-admission .

Therefore, necessary measures should be taken to diminish the intensity of PLSP. Although the exact mechanism of PLSP remains unclear, some studies have suggested that it is caused by the trapping of carbon dioxide (CO2) between the liver and the right diaphragm and subsequent conversion into carbonic acid, which irritates the diaphragm and subsequently generates referred shoulder pain (C4 dermatomal) . Therefore, several studies have attempted to decrease the incidence or severity of PLSP by promoting the removal of remaining CO2 from the abdominal cavity. These efforts include drainage tube insertion, intraperitoneal saline instillation (IPSI), and the usage of intraperitoneal local anesthetic agents . More-over, the pulmonary recruitment maneuver (PRM) can also facilitate the removal of CO2 from the abdominal cavity by increasing positive airway pressure and intrathoracic pressure. PRM is more commonly used in clinical practice because it does not require drugs, specialized apparatus, or additional medical costs, unlike the other methods . Several trials have described the advantages of PRM in patients undergoing laparoscopic operations compared to passive abdominal compression.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18- 65 years.

  * American Society of Anesthesiologists physical status classification (ASA) I - II
  * scheduled for an elective gyncologic laparoscopic procedures

Exclusion Criteria:

* • Urgent or emergency case.

  * ASA classification more than III.
  * Age less than 16 years.
  * Reduced left and right ventricular function (ejection fraction <40%).
  * Previous respiratory disease such as chronic obstructive pulmonary disease, restrictive lung disease, or had a history of thoracic or shoulder surgery
  * Patient conversion to a laparotomy.
  * the operation time is more than 3 h

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
post-laparoscopic shoulder pain by VAS score | 24 hours
  post-laparoscopic shoulder pain by VAS score

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Samarah BM, Shehada FA, Qaddumi J, Almasry NA, Alhroub N, ALBashtawy B, Mohammad K, ALBashtawy S, Alkhawaldeh A, ALBashtawy M, Al Omari O, Aljezawi M, Hamadneh S, Suliman M, Hani SB, ALBashtawy Z. The influence of the pulmonary recruitment maneuver on post-laparoscopic shoulder pain in patients having a laparoscopic cholecystectomy: a randomized controlled trial. Surg Endosc. 2023 Nov;37(11):8473-8482. doi: 10.1007/s00464-023-10450-x. Epub 2023 Sep 26. PMID 37752263
- [Background] Ryu KH, Lee SH, Cho EA, Kim JA, Lim GE, Song T. Comparison of impacts of intraperitoneal saline instillation with and without pulmonary recruitment maneuver on post-laparoscopic shoulder pain prevention: a randomized controlled trial. Surg Endosc. 2019 Mar;33(3):870-878. doi: 10.1007/s00464-018-6354-2. Epub 2018 Jul 16. PMID 30014331
- [Background] Demouron M, Selvy M, Dembinski J, Mauvais F, Cheynel N, Slim K, Sabbagh C, Regimbeau JM. Feasibility and Effectiveness of an Enhanced Recovery Program after Early Cholecystectomy for Acute Calculous Cholecystitis: A 2-Step Study. J Am Coll Surg. 2022 May 1;234(5):840-848. doi: 10.1097/XCS.0000000000000123. PMID 35426396